CLINICAL TRIAL: NCT02458118
Title: Study to Assess Pancreatic Blood Flow at Rest and During Stimulation Using Magnetic Resonance Imaging (fMRI) in Patients With Chronic Pancreatitis
Brief Title: Pancreatic Perfusion Using Secretin and MRI
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11109
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Pancreatitis
Keywords: chronic; pancreatitis; secretin; Blood flow
MeSH Terms: conditions — Pancreatitis, Chronic; Bronchiolitis Obliterans Syndrome; Pancreatitis | interventions — Secretin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Secretin (Experimental): Secretin 1 IU/kg over 3 min
  Interventions: Drug: Secretin

INTERVENTIONS:
Drug: Secretin — Secretin 1 IU/kg over 3 min
  Other Names: Secrelux" Sanochemia Pharmazeutika AG, Wein, Germany)

SUMMARY:
The purpose of this study is to assess pancreatic perfusion in patients with chronic pancreatitis at rest and after secretin stimulation and compare this to published data on pancreatic perfusion in normal subjects.

DETAILED DESCRIPTION:
Pancreatic blood flow or perfusion is difficult to quantify due to the complex vascular supply to the organ and its retroperitoneal location, adjacent to the abdominal aorta. The pancreas is supplied by the superior gastroduodenal artery from the celiac plexus, branches from the hepatic and splenic arteries, which originate from the celiac plexus, and the inferior gastroduodenal artery, which originates from the superior mesenteric artery. Identifying changes in flow in all these vessels with good spatial and temporal resolution is challenging but important in understanding many of the chronic conditions of the pancreas.

Chronic pancreatitis (CP) is an inflammatory condition of the pancreas leading to irreversible damage to the tissue. It is increasing in incidence in all nations, and is related to rising alcohol consumption and improved diagnostic techniques. In Europe the incidence is approximately 6-7/100,000 population. 73-91% of patients affected are male with an average age of 49-60yrs. Patients affected by CP have a high morbidity, such as diabetes and chronic abdominal and/or post-prandial pain in 80-90%, which required frequent hospital admission, control-drug prescriptions and intervention by specialist hospital services. However the mechanisms of chronic and post-prandial pain for CP patients are not well understood, but tissue ischaemia, inflammation and neurological changes have been proposed. These mechanisms may be inter-related with pancreatic inflammation and neurochemical changes, such as an increase substance P, which can produce vasoconstriction, reducing pancreatic perfusion and worsening ischaemia of intra-pancreatic nerves(3). A greater understanding of the ischaemic and inflammatory mechanisms behind the pain in CP, would greatly enhance the development of treatment for this and other debilitating conditions.

There are a few studies of pancreatic tissue perfusion in humans, those studies which have assessed perfusion have used invasive techniques such as endoscopic or laparoscopic measurement and hydrogen gas clearance methods. Although these methods have demonstrated decreased resting blood flow and little response to secretin stimulation in CP patients compared to healthy controls, the techniques are highly invasive, time consuming and expensive and can cause the participant significant morbidity. This has led to several non-invasive techniques including infusion of oxygen-15 water and positron emission tomography (PET), contrast-material-enhanced trans-abdominal ultrasound (US) or contrast-enhanced dynamic computer tomography (CT). However these techniques involve infusion of an exogenous marker to detect the change in flow rate and often require a radiation exposure or are operator dependant and give poor spatial or temporal resolution, limiting the usefulness of the studies.

MRI is an attractive alternative for the assessment of pancreatic perfusion, providing good spatial and temporal resolution with no radiation exposure. Two methods can be used, Contrast-Enhanced (CE) MRI or Arterial Spin Labelling (ASL) techniques. ASL provides a tool for quantitative assessment of tissue perfusion without the need for contrast administration.

Contrast-enhanced MRI using gadodiamide has been used to explore the changes in pancreatic perfusion with secretin stimulation. This study in 10 healthy volunteers demonstrated that at rest there was a higher blood flow within the body and the tail of the pancreas, compared to the head. With secretin stimulation there was a significant increased perfusion in all regions of the pancreas. ASL techniques, do not require exogenous contrast agents, only two previous studies have measured pancreatic perfusion with ASL, one exploring pancreatic exocrine functions in type 1 diabetics. A recent study at the Nottingham Digestive Diseases Centre on pancreatic perfusion measurement using ASL at baseline and after intravenous secretin stimulation has standardised the MRI technique of measuring pancreatic perfusion.

There are no studies using MRI ASL to measure pancreatic perfusion in patients with chronic pancreatitis after secretin stimulation. This pilot study aims to test the feasibility of using MRI ASL to measure pancreatic perfusion in patients with chronic pancreatitis with a view to perfecting the technique. This will allow future studies comparing pancreatic perfusion in healthy adult controls to patients with chronic pancreatitis thus improving the investigators understanding of the pathophysiology of pain in patients with chronic pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* Adults with chronic pancreatitis (as defined by the Cambridge criteria)

Exclusion Criteria:

1. Allergy to secretin
2. Claustraphobia
3. Refusal to consent for the study
4. MRI contraindications e.g. pacemaker, artificial heart valve
5. Previous abdominal surgery except appendectomy or hernia repair
6. History of chronic abdominal pain from causes other than pancreatitis eg. inflammatory bowel or coeliac disease
7. Pregnant women (safety concerns from injection of secretin)
8. Patients younger than 18 years of age

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-06; Primary Completion 2016-04 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Blood flow to pancreas as measured by arterial spin labelling MRI | 1.5 hours

SECONDARY OUTCOMES:
Change in blood flow to pancreas after intravenous secretin | 1.5 hours
Pancreatic diffusion | T 0, 5, 10, 20, 30, 40
Pancreatic volume | T 0, 5, 20, 40

CONTACTS AND LOCATIONS:
Overall Officials: John Simpson, Principal Investigator — University of Nottingham
Locations (1):
- 1.5T Brain and Body Imaging centre, University of Nottingham Campus, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andren-Sandberg A, Hoem D, Gislason H. Pain management in chronic pancreatitis. Eur J Gastroenterol Hepatol. 2002 Sep;14(9):957-70. doi: 10.1097/00042737-200209000-00006. No abstract available. PMID 12352215
- [Background] Jupp J, Fine D, Johnson CD. The epidemiology and socioeconomic impact of chronic pancreatitis. Best Pract Res Clin Gastroenterol. 2010 Jun;24(3):219-31. doi: 10.1016/j.bpg.2010.03.005. PMID 20510824
- [Background] Drewes AM, Krarup AL, Detlefsen S, Malmstrom ML, Dimcevski G, Funch-Jensen P. Pain in chronic pancreatitis: the role of neuropathic pain mechanisms. Gut. 2008 Nov;57(11):1616-27. doi: 10.1136/gut.2007.146621. Epub 2008 Jun 19. PMID 18566105
- [Background] Ceyhan GO, Demir IE, Maak M, Friess H. Fate of nerves in chronic pancreatitis: Neural remodeling and pancreatic neuropathy. Best Pract Res Clin Gastroenterol. 2010 Jun;24(3):311-22. doi: 10.1016/j.bpg.2010.03.001. PMID 20510831
- [Background] Lewis MP, Lo SK, Reber PU, Patel A, Gloor B, Todd KE, Toyama MT, Sherman S, Ashley SW, Reber HA. Endoscopic measurement of pancreatic tissue perfusion in patients with chronic pancreatitis and control patients. Gastrointest Endosc. 2000 Feb;51(2):195-9. doi: 10.1016/s0016-5107(00)70417-2. PMID 10650267
- [Background] Ishida H, Makino T, Kobayashi M, Tsuneoka K. Laparoscopic measurement of pancreatic blood flow. Endoscopy. 1983 May;15(3):107-10. doi: 10.1055/s-2007-1021480. PMID 6223807
- [Background] Kubo S, Yamamoto K, Magata Y, Iwasaki Y, Tamaki N, Yonekura Y, Konishi J. Assessment of pancreatic blood flow with positron emission tomography and oxygen-15 water. Ann Nucl Med. 1991 Nov;5(4):133-8. doi: 10.1007/BF03164627. PMID 1797067
- [Background] D'Onofrio M, Gallotti A, Principe F, Mucelli RP. Contrast-enhanced ultrasound of the pancreas. World J Radiol. 2010 Mar 28;2(3):97-102. doi: 10.4329/wjr.v2.i3.97. PMID 21160942
- [Background] Miles KA, Hayball MP, Dixon AK. Measurement of human pancreatic perfusion using dynamic computed tomography with perfusion imaging. Br J Radiol. 1995 May;68(809):471-5. doi: 10.1259/0007-1285-68-809-471. PMID 7788231
- [Background] Bali MA, Metens T, Denolin V, De Maertelaer V, Deviere J, Matos C. Pancreatic perfusion: noninvasive quantitative assessment with dynamic contrast-enhanced MR imaging without and with secretin stimulation in healthy volunteers--initial results. Radiology. 2008 Apr;247(1):115-21. doi: 10.1148/radiol.2471070685. Epub 2008 Feb 21. PMID 18292476
- [Background] Schraml C, Schwenzer NF, Martirosian P, Claussen CD, Schick F. Perfusion imaging of the pancreas using an arterial spin labeling technique. J Magn Reson Imaging. 2008 Dec;28(6):1459-65. doi: 10.1002/jmri.21564. PMID 19025955
- [Background] Hirshberg B, Qiu M, Cali AM, Sherwin R, Constable T, Calle RA, Tal MG. Pancreatic perfusion of healthy individuals and type 1 diabetic patients as assessed by magnetic resonance perfusion imaging. Diabetologia. 2009 Aug;52(8):1561-5. doi: 10.1007/s00125-009-1406-8. Epub 2009 Jun 3. PMID 19488737